CLINICAL TRIAL: NCT01791140
Title: Program for Assessment of Activity and Safety of 1st-line Bevacizumab (Avastin) Therapy in Elderly Patients With Metastatic Colorectal Cancer (BEVERLY-C Study)
Brief Title: BEVERLY-C: An Observational Study of Avastin (Bevacizumab) in First-Line Treatment in Elderly Patients With Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25630
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the efficacy and safety of Avastin (bevacizumab) in combination with fluoropyrimidine-based chemotherapy in elderly patients (>/= 65 years of age) with newly diagnosed metastatic colorectal cancer. Patients will be followed until disease progression, death, withdrawal of consent, discontinuation of physician-patient relationship or study closure, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 65 years of age
* Patients with newly diagnosed metastatic colorectal cancer starting first-line treatment with Avastin in combination with fluoropyrimidine-based chemotherapy according to the approved Hungarian Summary of Product Characteristics
* Patients suitable for Avastin treatment as assessed by the treating physician

Exclusion Criteria:

* Any contraindications to Avastin treatment according to the Hungarian Summary of Product Characteristics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (</= 65 years of age) with newly diagnosed metastatic colorectal cancer starting first-line treatment with Avastin in combination with fluoropyrimidine-based chemotherapy
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Median progression-free survival | approximately 3.5 years

SECONDARY OUTCOMES:
Overall response rate (complete response + partial response) | approximately 3.5 years
Clinical benefit rate (complete response + partial response + stable disease) | approximately 3.5 years
Metastasectomy rate | approximately 3.5 years
Mean duration of Avastin treatment | approximately 3.5 years
Safety: Incidence of adverse events | approximately 3.5 years
Median progression-free survival in subgroup receiving Avastin plus fluorouracil monotherapy | approximately 3.5 years
Median progression-free survival according to age group (65-74 years; >/= 75 years) | approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Budapest, Hungary